CLINICAL TRIAL: NCT00000861
Title: A Randomized Trial of Immediate Versus Deferred Indinavir in Addition to Background Antiretroviral Therapy in HIV-Infected Patients With CD4+ Cell Counts Between 200 and 500/mm3 and Plasma HIV RNA Levels >= 10,000 Copies/ml
Brief Title: The Addition of Indinavir to Anti-HIV Treatment in HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: CPCRA 041; 11591 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Administration Schedule; HIV Protease Inhibitors; CD4 Lymphocyte Count; Indinavir; RNA, Viral; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Indinavir

INTERVENTIONS:
Drug: Indinavir sulfate

SUMMARY:
The purpose of this study is to evaluate the effect of immediate versus deferred indinavir (IDV) in addition to background therapy on disease progression or death in patients with CD4+ cell counts between 200 and 500 cells/mm3 and plasma HIV RNA levels >= 10,000 copies/ml.

This study aims to examine two management strategies, immediate versus deferred IDV therapy, for their clinical effects in the context of background antiretroviral (AR) therapy, given according to current clinical practice. There is an urgent need to identify the optimal use of IDV in patient management, since clinical endpoint studies have not been completed in the United States. Since there is little information about the long term durability of clinical effects, and even less information about the timing of the initiation of protease inhibitor therapy, exploring the disease progression and survival impact of immediate versus delayed use of IDV will yield important information to guide clinical decision making for this group of patients.

DETAILED DESCRIPTION:
This study aims to examine two management strategies, immediate versus deferred IDV therapy, for their clinical effects in the context of background antiretroviral (AR) therapy, given according to current clinical practice. There is an urgent need to identify the optimal use of IDV in patient management, since clinical endpoint studies have not been completed in the United States. Since there is little information about the long term durability of clinical effects, and even less information about the timing of the initiation of protease inhibitor therapy, exploring the disease progression and survival impact of immediate versus delayed use of IDV will yield important information to guide clinical decision making for this group of patients.

Prior to randomization the patient and clinician will determine whether the background therapy will be zidovudine (ZDV) plus lamivudine (3TC) or other background antiretroviral therapy (OBAT). Patients will then be randomized to IDV or matching placebo. AS PER AMENDMENT 06/27/97: The protocol was closed as of 03/25/97, and all patients have been unblinded to their assigned treatment. Patients still on study medication are eligible for the protocol extension. Patients who were randomized to immediate IDV may continue on therapy for up to an additional 4 months. All study therapy, both for those on immediate or delayed therapy, must be discontinued on 10/24/97.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Topical and/or antifungal agents, except ketoconazole.
* Treatment, maintenance, or chemoprophylaxis with approved agents for OIs will be given as clinically indicated.
* Clinically indicated antibiotics, unless excluded.
* Systemic corticosteroid use for <21 days for acute problems is permitted as clinically indicated. However, chronic systemic corticosteroid use should be avoided.
* Recombinant erythropoietin (rEPO) and granulocyte-colony stimulating factor (G-CSF, filgrastim).
* Didanosine (ddI).
* Regularly prescribed medications, such as antipyretics, antidepressants, oral contraceptives, megestrol acetate, testosterone, or any other medication.

Patients must have:

* A working diagnosis of HIV infection.
* A CD4+ count between 200 and 500 cells/mm3.
* Signed, informed parental consent if patient is less than 18.

NOTE:

* The DAIDS Clinical Science Research Committee (CSRC) has deemed this protocol appropriate for prisoner enrollment.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following conditions or symptoms are excluded:

Febrile illness with temperature > 38.5 degrees C (101.3 degrees F) within 3 days prior to study entry.

Concurrent Medication:

Excluded:

* Non-nucleoside reverse transcriptase inhibitors.
* Protease inhibitors except IDV.
* Rifabutin and rifampin.
* Ketoconazole.
* Terfenadine, astemizole, cisapride, triazolam and midazolam.

Patients with any of the following prior conditions are excluded:

* History of prior saquinavir (SQV) therapy for more than 14 days.
* History of any prior protease inhibitor therapy other than SQV.
* History of serious opportunistic infection.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1900
Dates: Study Completion 1997-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saravolatz L, Study Chair; Crane L, Study Chair; Mayers D, Study Chair
Locations (14):
- United States (14):
  - Community Consortium of San Francisco, San Francisco, California
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Veterans Administration Med Ctr / Regional AIDS Program, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Comprehensive AIDS Alliance of Detroit, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - Southern New Jersey AIDS Cln Trials / Dept of Med, Camden, New Jersey
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Richmond AIDS Consortium, Richmond, Virginia

REFERENCES:
- [Background] Spector SA, Barker C, Buhles W, Feinberg J, Montague P, Weingeist T, DeArmond B. A randomized, controlled study of immediate vs deferred ganciclovir therapy in AIDS patients with cytomegalovirus peripheral retinitis. Int Conf AIDS. 1991 Jun 16-21;7(1):44 (abstract no MB86)